CLINICAL TRIAL: NCT04800874
Title: An Open Label Phase 2 Study of BBP-418 in Patients With Limb Girdle Muscular Dystrophy Type 2I (MLB-01-003)
Brief Title: Study of BBP-418 in Patients With LGMD2I
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ML Bio Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MLB-01-003
Record Dates: First submitted 2021-01-25; First posted 2021-03-16 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: LGMD2I
Keywords: LGMD; LGMD R9; Limb Girdle Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Limb-Girdle, Type 2I; Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Intervention Model Description: Subjects must have been enrolled in the MLB-01-001 study to participate in this trial. Three ascending dose cohorts of 4-6 subjects each are planned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Subjects will receive 6 grams of BBP-418 once daily x 90 days, then 12 grams twice daily (BID, a least 8 hours apart) of BBP-418 daily until study completion.
  Interventions: Drug: BBP-418
- Cohort 2 (Experimental): Subjects will receive 6 grams of BBP-418 twice daily (BID, at least 8 hours apart) x 90 days, then 12 grams BID of BBP-418 daily until study completion.
  Interventions: Drug: BBP-418
- Cohort 3 (Experimental): Subjects will receive 12 grams of BBP-418 twice daily (BID, at least 8 hours apart) x 90 days, then 12 grams BID of BBP-418 daily until study completion.
  Interventions: Drug: BBP-418

INTERVENTIONS:
Drug: BBP-418 — BBP-418 is being developed for the treatment of patients with Limb-Girdle Muscular Dystrophy Type 2I (LGMD2I) for which no approved therapy currently exists. It targets the molecular defect at the source by supplying excess substrate to the mutant enzyme thus boosting glycosylation of muscle α-dystroglycan. The BBP-418 drug product will be packaged in sachets and provided in a carton for in-clinic and at home use.

SUMMARY:
BBP-418 is being developed for the treatment of patients with Limb-Girdle Muscular Dystrophy Type 2I (LGMD2I). This is an open label study to determine the safety and tolerability of ascending dose levels of BBP-418 in the treatment of ambulatory and non-ambulatory patients with LGMD2I for which no approved therapy currently exists.

DETAILED DESCRIPTION:
This is an open label study in ambulatory and non-ambulatory subjects with LGMD2I (also known as LGMD R9) previously enrolled in the natural history Study MLB-01-001. This is a study to determine the safety and tolerability of ascending dose levels of BBP-418 in those subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have a body weight >30 kg
* Have a genetically confirmed diagnosis of LGMD2I and be clinically affected (defined as demonstrating clinical weakness on bedside evaluation in either a limb-girdle pattern, or in a distal extremity)
* Able to complete the 10-meter walk test in ≤ 12 seconds unaided ("moderate disease") or are with "severe disease"/non-ambulatory as defined by being unable to complete the 10-meter walk unaided in >12 seconds
* Willing to use an adequate method of contraception from time of consent through 12 weeks after last dose
* Previous enrolment in the Natural History study MLB-01-001

Exclusion Criteria:

* Evidence of clinically significant concomitant disease, including:

  * Any history of a gastrointestinal condition, including surgeries, which may affect absorption after oral administration
  * Any significant concomitant medical condition, including cardiac, pulmonary, renal, hepatic or endocrine disease other than that associated with LGMD2I
  * Any condition other than LGMD2I requiring therapy with prescription medicine (medication for common and mild concomitant conditions may be permitted after consultation with the PI)
  * Any other laboratory, vital sign, ECG abnormality, or clinical history or finding that, in the investigator's opinion, is likely to unfavorably alter the risk-benefit of study participation, confound study results, or interfere with study conduct or compliance
* If pregnant and/or breastfeeding or planning to conceive children within the projected duration of the study through 12 weeks after the last dose of study treatment.
* History of drug abuse including alcoholism within 2 years prior to consenting
* Use of ribose or other sugar alcohol-containing supplement within 60 days of Day 1
* Use of a corticosteroid within 60 days of Day 1
* Presence of a platelet disorder, bleeding disorder or other contraindication to muscle biopsy
* Actively on an experimental therapy or device or was on an experimental therapy or device within 60 days prior to Day 1.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) that lead to dose decrease or discontinuation | 60 months

SECONDARY OUTCOMES:
Pharmacokinetic profile of BBP-418 by assessment of maximum concentration (Cmax) | 24 months
Changes in pharmacodynamic parameters by assessing changes in levels of N-terminal fragment of alpha dystroglycan (α-DG) | 24 months
Changes in pharmacodynamic parameters by assessing muscle biopsy of the tibialis anterior | 24 months
Pharmacokinetic profile of BBP-418 by assessment of area under the curve (AUC) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy Harper, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No